CLINICAL TRIAL: NCT05129631
Title: HEARTPrep: A Virtually-delivered Psychosocial Intervention for Mothers Expecting a Baby With Congenital Heart Disease
Acronym: HEARTPrep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Erica Sood, Pediatric Psychologist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1813613
Record Dates: First submitted 2021-10-31; First posted 2021-11-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEARTPrep (Experimental): HEARTPrep is a virtually-delivered psychosocial intervention for mothers expecting a baby with CHD. HEARTPrep consists of three distinct modules: Adjusting, Connecting, and Preparing. Each module targets one distinct primary outcome (emotional distress, social isolation, parenting self-efficacy) and a common secondary outcome (hope) through a suite of evidence-based intervention elements (e.g., psychoeducation, cognitive restructuring, mindfulness) for addressing emotional problems in other populations, including pregnant women. HEARTPrep elements include: a) telehealth with a psychosocial provider, b) recorded videos, c) educational tools, and d) links to resources.
  Interventions: Behavioral: HEARTPrep

INTERVENTIONS:
Behavioral: HEARTPrep — HEARTPrep is a virtually-delivered psychosocial intervention for mothers expecting a baby with CHD.

SUMMARY:
Congenital heart disease (CHD) is the most common birth defect and is increasingly diagnosed prenatally. Mothers describe their prenatal experiences as highly stressful and traumatic after a diagnosis of CHD. Maternal stress during pregnancy exerts a powerful influence on birth outcomes and developmental trajectories, particularly for children in underserved populations. In partnership with diverse parent and clinician stakeholders, our team designed HEARTPrep, an innovative, virtually-delivered psychosocial intervention for mothers expecting a baby with CHD. This project will pilot HEARTPrep with mothers expecting a baby with CHD to obtain preliminary data for a larger future trial. This intervention has the potential to improve emotional wellbeing in mothers expecting a baby with CHD, thereby altering developmental trajectories for this large population of children.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most common birth defect and is increasingly diagnosed prenatally. Mothers describe their prenatal experiences as highly stressful and traumatic after a diagnosis of CHD. Maternal stress during pregnancy exerts a powerful influence on birth outcomes and developmental trajectories, particularly for children in underserved populations. Targeted efforts to mitigate impacts of maternal stress for this highly vulnerable population are lacking. In partnership with diverse parent and clinician stakeholders, the investigators designed HEARTPrep, an innovative, virtually-delivered psychosocial intervention for mothers expecting a baby with CHD. HEARTPrep will be delivered through the Nemours App, an accessible tool for telehealth and patient education. The investigators aim to determine whether HEARTPrep modules produce clinically significant improvements on outcomes in mothers expecting a baby with CHD (Proof-of-Concept). This program of research has the potential to improve emotional wellbeing in mothers expecting a baby with CHD, thereby altering developmental trajectories for this large population of children.

ELIGIBILITY:
Inclusion Criteria:

* Expectant mothers carrying a fetus with congenital heart disease expected to require cardiac surgery in the first year of life
* Partners of participating expectant mothers can also participate together with the mother
* Receiving fetal cardiac care at Nemours Children's Health
* Speaks English or Spanish fluently
* Age 18 or older
* Access to a computer, tablet or mobile device with internet access

Exclusion Criteria:

-Fetus has a genetic syndrome or other comorbid condition associated with a life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
HEARTPrep Evaluation Questionnaire | Post-intervention
  Assesses perceived acceptability and feasibility of HEARTPrep (item responses range from 0-4 with higher scores reflecting greater acceptability and feasibility; minimum score = 0; maximum score = 64)
Change in Emotional Distress - Patient-Reported Outcomes Measurement Information System (PROMIS) Short-Form | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assesses change from baseline in feelings of anxiety and depression (item responses range from 1-5 with higher scores reflecting greater emotional distress; minimum score = 4; maximum score = 20)
Change in Social Isolation - PROMIS Short-Form | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assesses change from baseline in feelings of social isolation (item responses range from 1-5 with higher scores reflecting greater social isolation; minimum score = 4; maximum score = 20)
Change in Parenting Self-Efficacy - PROMIS Short-Form | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assesses change from baseline in feelings of parenting self-efficacy (item responses range from 1-5 with lower scores reflecting lower parenting self-efficacy; minimum score = 4; maximum score = 20)

SECONDARY OUTCOMES:
Change in Hope - PROMIS Short-Form | Weeks 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
  Assesses change from baseline in feelings of hope (item responses range from 1-5 with lower scores reflecting lower hope; minimum score = 4; maximum score = 20)

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States